CLINICAL TRIAL: NCT03887000
Title: Effect of Magnesium on Stress in Fibromyalgia: Randomized Double-blind Placebo Controlled Trial
Brief Title: Magnesium, Stress and Fibromyalgia
Acronym: SeMAFor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: CIC Inserm 1405, University Hospital Clermont-Ferrand, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHU-429; 2018-A02059-46 (Other: 2018-A02059-46)
Record Dates: First submitted 2019-03-07; First posted 2019-03-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Stress; Magnesium; Sleep disorders
MeSH Terms: conditions — Fibromyalgia; Sleep Wake Disorders | interventions — Magnesium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAGNESIUM (Experimental): Fibromyalgia patients taking either magnesium or placebo according to the randomized plan
  Interventions: Other: magnesium; Other: placebo
- PLACEBO (Experimental): Fibromyalgia patients taking either magnesium or placebo according to the randomized plan
  Interventions: Other: magnesium; Other: placebo

INTERVENTIONS:
Other: magnesium — Fibromyalgia patients taking either magnesium or placebo according to the randomized plan
Other: placebo — Fibromyalgia patients taking either magnesium or placebo according to the randomized plan

SUMMARY:
Fibromyalgia affects an average of 2% of the French population. Data from the literature report that low levels of magnesium could be associated with fibromyalgia. However, no study to date has investigated the effect of oral magnesium administration on stress in fibromyalgia.

This trial therefore aims to evaluate whether magnesium could improve stress and the various disorders that contribute to the complexity of fibromyalgia, including pain, cognition, sleep disorders and quality of life.

DETAILED DESCRIPTION:
This is an interventional, randomized, placebo-controlled, double blind study of the use of magnesium in fibromyalgia. The effect of magnesium on stress measured by DASS-42 over 28 days after taking magnesium / placebo will be studied.

The secondary objectives will evaluate the evolution of the scores of all the tests and questionnaires carried out before taking magnesium or placebo (D0: Visit 2), then at D0 + 28 (visit 3) and D0 + 84 days (visit 4 corresponding to the end-of-study visit).

Secondary parameters are the following :

Impact of fibromyalgia, heart rate variability, pain intensity, cognition, feelings of patients, impression of change, sleep quality, fatigue intensity, social vulnerability, catastrophism, presence of small fiber neuropathy, stress induced by colors, pain induced by thermal stimulation, concentration of magnesium, analysis of microbiota and evaluation of genetic factor.

Blood magnesium and magnesuria will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18,
* Patient with fibromyalgia according to the criteria of the 2016 ACR,
* Patient presenting a score on the DASS-42 > 18 scale,
* Patient free from any initiation of new treatment or diet at the time of inclusion,
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Acceptance to give written consent,
* Affiliation to the French Social Security system,
* Registration or acceptance of registration in the National Register of Volunteers participating in research.

Exclusion Criteria:

* having a contraindication to the administration of magnesium: hypersensitivity to magnesium chloride, or to any of the excipients,
* with a magnesium concentration of > 1.05 mmol / l,- with severe renal impairment with a creatinine clearance < 30 ml / min,
* receiving a treatment or dietary supplement containing magnesium at the time of inclusion,
* treated with antibiotics in the three months prior to inclusion,- who has reported gastroenteritis in the two months prior to inclusion,
* physically unfit to place the palms or soles of the feet on the Sudoscan® electrodes,
* having a medical and / or surgical history judged by the investigator or his representative to be incompatible with the test (in particular a disease known to cause small fiber neuropathies: diabetes, Sjögren's disease, vasculitis, sarcoidosis, chronic ethylism ....),
* using anticoagulant therapy or allergy to local anesthetics,- of childbearing age not using an effective contraceptive method, pregnant or breastfeeding woman.
* participating in another clinical trial, or being in the exclusion period, or having received a total amount of benefits exceeding EUR 4500 over the 12 months preceding the start of the trial,
* having cooperation and understanding that does not allow strict compliance with the conditions laid down in the Protocol,
* benefiting from a measure of legal protection (guardianship, guardianship, deprivation of liberty, safeguard of justice),
* not affiliated to the French Social Security system.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Measure of stress with DASS-42 | at day 0
  Measure of stress with stress subscale in magnesium and placebo group. This subscale consists of 14 questions of self-evaluation

SECONDARY OUTCOMES:
Evaluation of the impact of fibromyalgia using the FIQ questionnaire | Day0; Day0+28; Day0+84
  The revised FIQ questionnaire is a 10-item self-questionnaire that assesses the impact of fibromyalgia
Detection of fibromyalgia using the FIRST questionnaire | Day0; Day0+28; Day0+84
  The FIRST questionnaire is a 6-item self-questionnaire that detects fibromyalgia.
Evaluation of stress by the heart rate variability | Day0-7; Day0; Day0+28; Day0+84
  Heart rate variability (HRV / HRV) is a measure of changes in heart rate that will provide an estimate of stress. It is usually calculated by analyzing time series of beat-by-beat intervals of the ECG or blood pressure plots.
Assessment Using Numerical Scale (EN) | Day0; Day0+28; Day0+84
  This scale allows the patient to note the pain on a graduation whose minimum score is 0 and the maximum score is 10.
Concise Pain Questionnaire (QCD) | Day0; Day0+28; Day0+84
  This self-assessment scale allows the patient to characterize the pain in relation to its psychosocial intensity and impact. The patient is asked to answer 9 graduated questions by circling a number from 0 (no pain) to 10 (the most horrible pain you can imagine).
Evaluation of the impact on cognition by the Trail Making Test A and B (TMT A and B) and the Cantab® test | Day0; Day0+28; Day0+84
  The Trail Making Test (TMT) is recognized as one of the most frequently used neuropsychological tests in clinical practice alternating numbers and letters (1-A-2-B-3- C, etc.).
  The Cantab® is a comprehension test, executive functions, memory, attention and decision-making.
Evaluation of the impact on cognition by the Trail Making Test A and B (TMT A and B) | Day0; Day0+28; Day0+84
  The Trail Making Test (TMT) is recognized as one of the most frequently used neuropsychological tests in clinical practice alternating numbers and letters (1-A-2-B-3- C, etc.).
Cantab® test | Day0; Day0+28; Day0+84
  The Cantab® is a comprehension test, executive functions, memory, attention and decision-making.
Evaluation of the emotions by visualization of images and scale evaluating the feelings of the patients | Day0; Day0+28; Day0+84
  The International Affective Picture System (IAPS) is a library of 1200 standardized images that can induce an emotional reaction, constituting as many emotional stimuli (positive or negative) or not (neutral).
Evaluation of the overall impression of change by the Patient Global Impression of Change Questionnaire (PGIC) | Day0; Day0+28; Day0+84
  The Global Impression of Change Patient is a scale of global perception of change ("deterioration" or "improvement") completed by the patient. This scale is graduated from 1 = much better to 7 = significantly worse
Evaluation of the impact on the Pittsburg Sleep Quality Index (PSQI) | Day0; Day0+28; Day0+84
  The Pittsburg Sleep Quality Index is a self-administered questionnaire with 19 items. It has been developed to measure the quality of sleep in the month preceding the interview with the patient. This questionnaire has 7 components: subjective sleep quality, sleep latency, sleep duration, usual sleep efficiency, sleep disorders, use of a sleep medication, and poor daytime fitness
Evaluation of the intensity of fatigue by the Fatigue Severity Scale (FSS) | Day0; Day0+28; Day0+84
  The fatigue severity scale is a 9-item self-questionnaire to assess the patient's fatigue intensity. The patient is asked to circle a number from 1 to 7 for each question, a low value representing a low intensity
Social Vulnerability Assessment (EPICES) | Day0; Day0+28; Day0+84
  The EPICES questionnaire is composed of 11 binary questions (yes / no) allowing to calculate an individual score indicating the precariousness and inequalities of health ranging from 0 to 100.
Evaluation of catastrophism by the PCS (Pain Catastrophizing Scale) scale | Day0; Day0+28; Day0+84
  Pain Catastrophizing Scale (PCS) is a questionnaire in which the patient is asked to describe the kind of thought and emotions they feel during pain. This questionnaire consists of 13 items describing different thoughts or emotions that may be associated with the pain. The patient will have to indicate how much he has these thoughts or emotions when he feels pain by giving a score between 0 and 4, 0: not at all, 4: all the time. The final score is the sum of the scores for each question.
Quality of life (Short Form 12 items Short Form survey) | Day0; Day0+28; Day0+84
  assessed by a quality of life questionnaire (Short Form 12 items Short Form survey (SF12)
Evaluation of the presence of small fiber neuropathy (Sudoscan® ) | AT Day0; Day0+28
  Sudoscan® (Impeto Medical, Paris, France) is a new device that provides a rapid, non-invasive and reproducible quantitative assessment of sweat function.
Evaluation of the presence of small fiber neuropathy (skin biopsy) | at Day0
  A skin biopsy will be realized for histological analysis to determine the presence of small fiber neuropathy.
plasma magnesium dosage | D0; D0+28; D0+84
  The intracellular magnesium concentrations will be determined by the blood samples taken at the inclusion visit, at the end of the treatment on visit 3 (D0 + 28) and on visit 4 (D0 + 84).
erythrocyte magnesium dosage | D0; D0+28; D0+84
  The erythrocyte magnesium concentrations will be determined by the blood samples taken at the inclusion visit, at the end of the treatment on visit 3 (D0 + 28) and on visit 4 (D0 + 84).
urinary magnesium dosage | D0; D0+28; D0+84
  The urinary concentration of magnesium will be determined by the urine collected for 24 hours, the day before visits 3 and 4.
urinary magnesium dosage | D0+28; D0+84
  The urinary concentration of magnesium will be determined by the urine collected for 24 hours, the day before visits 3 and 4.
creatinine dosage | D0-7
  The creatinine concentrations will be determined by the blood samples taken at the inclusion visit.
Analysis of the microbiota (stool samples) | 24 hours before the visit 2
  Analysis of the microbiota: the patient must carry out the collection at her home maximum 24 hours before the visit 2 by following the technical instructions described in the explanatory note that will be provided. She will then ensure that the stool preservation and transport procedure described in this document is followed.
Evaluation of genetic polymorphism using OpenArray technology | Day0-7
  Identification of genes involved
Evaluation of stress response during visual stimulation | Day0; Day0+28
  Stress intensity will be assessed by the numerical stress rating scale: the scale ranges from 0 "no stress" to 10 "maximal stress" following different visual stimulation induced by different colors during the anticipatory phase of pain.
Evaluation of pain response during thermal stimulation | Day0; Day0+28
  Pain intensity will be assessed by the numerical pain rating scale (NPRS): the scale ranges from 0 "no pain" to 10 "maximal tolerable pain" following different thermal stimulations (using Pathway Medoc®).
Evaluation of electromyography (EMG) of median nerve | day 0
  EMG motor and sensitive of the median nerve on both arm to control the speed of electrical conduction. For this purpose, we will measure the amplitude, latency and speed for the motor test, and the amplitude and speed for the sensitivity test.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France